CLINICAL TRIAL: NCT07404254
Title: A Randomized, Double-Blind, Parallel Trial to Assess Subjective and Physiological Responses to Consumption of Caffeinated Beverages in Healthy Adults With a Caffeine Routine
Brief Title: Effects of Variations in Caffeinated Beverages on Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GUAYAKI SUSTAINABLE RAINFOREST PRODUCTS, INC. (Industry)
Collaborators: Nlumn LLC (Unknown); Alethios, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NL-2503
Record Dates: First submitted 2026-01-12; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Caffeine; Beverage Intake
Keywords: caffeine beverages in health and well-being

STUDY DESIGN:
Intervention Model Description: This interventional trial focuses on evaluating the effects of the intervention on health and well-being.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeinated, low sugar beverage (Active Comparator)
  Interventions: Other: Caffeinated, low sugar beverage
- Caffeinated beverage (Active Comparator)
  Interventions: Other: Caffeinated beverage
- Control beverage (Placebo Comparator)
  Interventions: Other: Control beverage

INTERVENTIONS:
Other: Caffeinated, low sugar beverage — Participants will consume a caffeinated beverage with variations in sweetener and caffeine content.
  Arms: Caffeinated, low sugar beverage
Other: Caffeinated beverage — Participants will consume a caffeinated beverage with variations in sweetener and caffeine content.
  Arms: Caffeinated beverage
Other: Control beverage — Participants will consume a caffeinated beverage with the control level of sweetener and caffeine content.
  Arms: Control beverage

SUMMARY:
This study will evaluate post-beverage subjective caffeine responses and physiological responses to caffeinated beverage variations in generally healthy adults.

DETAILED DESCRIPTION:
This will evaluate post-beverage subjective caffeine responses using visual analog scale questionnaires, mood, quality of life, and physiological responses to ingredient variations in caffeine beverages.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥18 to ≤55 years of age
2. BMI ≥18.5 and <35.0 kg/m2
3. Generally good health
4. Participant currently and consistently has a sweetened caffeine routine
5. Participant is willing to substitute their current caffeine routine for the test beverage daily
6. Participant has never consumed the test beverage or similar products
7. Participant currently owns a wearable and is willing to use and connect the wearable device
8. Willing to use personal smart phone, tablet, or personal computer with stable internet connection
9. Willing and able to comply with all study procedures
10. Willing to adhere to all study procedures, including lifestyle considerations and sign forms providing informed consent to participate in the study

Exclusion Criteria:

1. History or presence, on the basis of the health history, of clinically important condition or disease states
2. Is currently following, or planning to be on, a weight loss regimen
3. Weight loss or gain >4.5 kg
4. History of gastrointestinal surgery for weight reducing purposes or gastrointestinal (GI) conditions
5. History of an eating disorder (e.g., anorexia nervosa or bulimia nervosa, binge eating) at the discretion of the Clinical Investigator.
6. History of unconventional sleep patterns (e.g., night shift) or diagnosed sleep disorder
7. Use of tobacco/nicotine products
8. Use of hemp/marijuana products
9. Unstable use of any prescription medication
10. Use of any medications(s) or dietary supplement(s), containing caffeine, or interacting with caffeine
11. Recent history of alcohol or substance abuse
12. Exposed to any non-registered drug product
13. Self-report of hypertension/high blood pressure without use of hypertensive medications
14. Any known allergy or intolerance to any ingredients contained in the study product
15. Any signs or symptoms of active infection of clinical relevance
16. History or presence of cancer, except for non-melanoma skin cancer
17. History of any major trauma or major surgical event
18. Female who is pregnant, planning to be pregnant during the study period, lactating
19. An employee, close relative of an employee, or participant who has a financial interest in Sponsor company or any other caffeine beverage company.
20. Any condition the Investigator believes would interfere with the participant's ability to provide informed consent or comply with the study protocol
21. A clinically significant medical condition that is affected by caffeine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Subjective caffeine visual analog scales | Day 5
  Participants will rate how they feel on a horizontal line. Lines will be flanked with perceived feelings. Scores range from 0-100, where a higher score indicates increase in that feeling.

SECONDARY OUTCOMES:
Subjective caffeine visual analog scales | Up to 5 hours after beverage consumption
  Participants will rate how they feel on a horizontal line. Lines will be flanked with perceived feelings. Scores range from 0-100, where a higher score indicates increase in that feeling.
Subjective quality of life ratings | Day 5
  Participants will rate how they feel using a Likert scale from 0-5. Where higher score indicate higher frequency in that feeling.
Physiological response - Sleep | Up to 5 hours post-beverage consumption and after 5 days of daily beverage consumption
  Sleep time in hours will be collected on wearable-derived algorithms (Apple Health, Garmin, or Fitbit).
Physiological responses - Activity | Up to 5 hours post-beverage consumption and after 5 days of daily beverage consumption
  Activity in step count will be collected on wearables (Apple Health, Garmin, or Fitbit) via accelerometry.

OTHER OUTCOMES:
Physiological responses - Heart rate | Up to 5 hours post-beverage consumption and after 5 days of daily beverage consumption
  Data collected by wearables
Subjective beverage experience ratings | Day 5
  Participants will rate how they feel on a horizontal line. Lines will be flanked with perceived feelings. Scores range from 0-100, where a higher score indicates increase in that feeling.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Nieman, PhD, Principal Investigator — Nlumn LLC
Locations (1):
- Alethios, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No